CLINICAL TRIAL: NCT04739579
Title: Post-operative CRP Trend May Lead to Early Diagnosis of Anastomotic Leak After Ileocolic Resection in Crohn's Disease Patients.
Brief Title: Post-operative CRP Trend After Ileocolic Resection in Crohn's Disease Patients.
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, ADELINE GERMAIN, Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI287
Record Dates: First submitted 2021-01-28; First posted 2021-02-04 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Anastomotic Leak; C-Reactive Protein
MeSH Terms: conditions — Crohn Disease; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anastomotic Leak
  Interventions: Diagnostic Test: C-Reactive Protein
- Non-Anatomotic Leak
  Interventions: Diagnostic Test: C-Reactive Protein

INTERVENTIONS:
Diagnostic Test: C-Reactive Protein — C-Reactive Protein trend in post-operative course

SUMMARY:
Our aim is to analyze C-Reactive Protein trends during the post-operative course in Crohn's Disease patients having undergone ileocolic resection and primary anastomosis, for the purpose of anastomotic leak early diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease patients
* Primary ileocolic anastomosis
* C-Reactive Protein data available in medical file

Exclusion Criteria:

* Protective stoma
* Associated resection with or without anastomosis during intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ileocolic resection with primary anastomosis
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak | up to 30 days following surgery
  Presence of a collection in the area of the anastomosis on computed tomography scan or evident anastomotic dehiscence at reoperation for peritonitis.

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Germain, MD, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU de Nancy, Nancy, France